CLINICAL TRIAL: NCT00937443
Title: Effectiveness of a Walking Program Modulating Cardioreparative Factors in Heart Failure
Acronym: EPCCHFWalk
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Vanderbilt_University
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure
Keywords: Physical Activity; Cardiac Heart Failure; Exercise Regimen; Cardioreparative Factors
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Physical Fitness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 60 ml of blood will be used to measure baseline levels of EPC's, NRG-1, VEGF, and SDF-1. Repeat venipuncture will be done at Week 12. Approximately 60 ml of blood for the measurement of EPC's, NRG1, VEGF, and SDF-1.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Walking Exercise Group: Walking Exercise Group versus Control Group
  Interventions: Other: Physical Fitness; Biological: Walking Exercise Group

INTERVENTIONS:
Other: Physical Fitness — Does intensity of aerobic walking exercise modify cardiac reparative factors
  Other Names: Quality of Life Questionnaires
Biological: Walking Exercise Group — Walking Group will increase intensity, duration, and steps of walking per week.
  Other Names: Quality of Life Questionnaires

SUMMARY:
The incidence of heart failure grows as the population continues to age. Heart failure incidence approaches 10 per 1,000 persons after the age of 65. Although pharmacotherapy improves the treatment of heart failure it remains insufficient in preventing the progression of this debilitating disease. Cell based therapy has gained great strides over the last decade, launching cellular therapy into the mix of artillery for the treatment of chronic heart failure and coronary disease. While early pre-clinical work demonstrates that stem cell based therapy improves heart failure the exact mechanism in which these endothelial progenitor cells (EPC's) are recruited from the bone marrow, proliferate under the mediation of growth factors, and migrate to the injured tissues endogenously still remains obscured. Therefore in order for clinicians and scientist to impact heart failure treatment, a greater understanding of the physiological changes in EPC's and other modulators of cardioreparative process need further investigation.

DETAILED DESCRIPTION:
Heart failure remains a devastating progressive chronic disease in which pharmacotherapy is not often sufficient. Although cell based therapy is gaining publicity in the treatment of coronary artery disease and heart failure. Determining how endothelial progenitor cells are recruited, proliferate, and home to injured tissue is an important area of investigation. Equally important is determining factors which improve EPC stimulation and efficiency such as realistic levels of exercise and the modulation of various cardioreparative factors (VEGF, NRG-1, and SDF-1) within heart failure patients. Since the endogenous repair mechanism is down regulated in heart failure patients such efforts may uncover ways to tip the balance in heart failure back to normal reparative maintenance.

ELIGIBILITY:
Inclusion criteria:

1. Subjects 30-65 years old.
2. Subjects able to give Informed Consent.
3. Subjects who will give permission for collection of clinical and demographic data from the electronic medical records.
4. Subjects with symptomatic ischemic or non-ischemic heart failure in a stable condition with New York Heart Association class II-III for at least the last 3 months before study enrollment.

   * Left ventricular ejection fraction (LVEF) < 40%.
   * Peak volume of oxygen utilization (peak VO2) of < 25 ml/kg/min.
5. Patient on a stable dose of statin or who can be initiated on statin therapy.
6. Subjects with ischemic cardiomyopathy must have had either a negative stress test within the last 6 months or a cardiac catheterization within the last year confirming stable disease.

Exclusion criteria:

1. Subjects with myocardial infarction or unstable angina within the last six months.
2. Subjects with symptomatic or severe aortic stenosis.
3. Subjects with severe HTN (SBP > 180) or hypotension (SBP < 100).
4. Subjects who are pregnant.
5. Subjects who have bone marrow suppression.
6. Subjects with exercise limiting peripheral arterial disease.
7. Subjects with history of ventricular tachycardia without an implantable defibrillator
8. Subjects with decompensated diabetes (HgA1c >10).
9. Subjects with orthopedic limitations.
10. Subjects with any other clinical condition precluding regular participation in walking exercise regimen.
11. Subjects who already participate in regular physical exercise regimen for greater than 30 minutes a day 5 days per week.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac Heart Failure Patients
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
endothelial progenitor cells | 12 Weeks

SECONDARY OUTCOMES:
exercise | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B Saywer, MD, PhD, Study Director — Vanderbilt Heart and Vascular Institute
Locations (1):
- Vanderbilt Heart and Vascular Institute, Nashville, Tennessee, United States